CLINICAL TRIAL: NCT02009969
Title: Serial Comparisons of Abdominal and Neurological MRI Scans of Patients With Refractory Psychosis Disorders
Brief Title: Serial Comparisons of Abdominal and Neurological MRI Scans
Acronym: SCANMRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H13-01685
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Psychotic Disorders
Keywords: Psychosis; Adverse effects; Symptom Severity; Magnetic Resonance Imaging
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare abdominal weight gain and fat distribution to changes in brain morphology in people taking antipsychotic medications.

DETAILED DESCRIPTION:
Abdominal weight gain is a significant side effect of antipsychotic medications. It has even been suggested to be part of the pathology of severe mental illnesses. Studies have shown that in persons with bipolar disorder, increased body mass index (BMI) is associated with irregular changes in the brain. This association has not been tested in persons with psychosis. In this study, we will be measuring abdominal fat distribution as measured by MRI to see if this is associated with abnormal brain morphology.

ELIGIBILITY:
Inclusion Criteria:

* Must be admitted to the BC (British Columbia) Psychosis Program at UBC (University of British Columbia) Hospital
* Must have clinically diagnosed psychosis (e.g. schizophrenia)
* Must be fluent in English
* Must not be contraindicated for MRI (i.e., must not be claustrophobic, have metal in the body, be pregnant, have BMI greater than or equal to 40, etc.)

Exclusion Criteria:

• None, other than those listed above

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have recently been seen at the BC (British Columbia) Psychosis Program at the University of British Columbia hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Abdominal distribution of visceral fat versus subcutaneous fat | Baseline (within 2 weeks of admission), 12 weeks later, and prior to discharge
  Change over time in amounts of visceral and subcutaneous fat as measured by automated segmentation of a magnetic resonance image (MRI)
Changes in total brain volume | Baseline (within 2 weeks of admission), 12 weeks later, and prior to discharge
  Change over time in total brain volume as measured by automated segmentation of a magnetic resonance image (MRI).
Changes in grey matter volume in the brain | Baseline (within 2 weeks of admission), 12 weeks later, and prior to discharge
  Change over time in amounts of brain grey matter as measured by automated segmentation of a magnetic resonance image (MRI).
Changes in white matter volume in the brain | Baseline (within 2 weeks of admission), 12 weeks later, and prior to discharge
  Change over time in amounts of brain white matter as measured by automated segmentation of a magnetic resonance image (MRI).
Changes in the volume of brain structures | Baseline (within 2 weeks of admission), 12 weeks later, and prior to discharge
  Change over time in the volume of brain structures as measured by automated segmentation of a magnetic resonance image (MRI).

SECONDARY OUTCOMES:
Comparing changes in abdominal fat distribution/accumulation to psychosis symptom severity | Baseline (within 2 weeks of admission), 12 weeks later, and prior to discharge
  To determine if an association exists between abdominal fat accumulation/distribution and psychosis symptom severity, as measured by the amounts of visceral and subcutaneous fat by automated segmentation of a magnetic resonance image (MRI) and standardized symptom rating scales, cognitive tests, and other neuropsychological examinations, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair M Barr, Ph.D., Principal Investigator — The University of British Columbia
Locations (1):
- BC Mental Health & Addictions Research Institute, Vancouver, British Columbia, Canada